CLINICAL TRIAL: NCT01243060
Title: Effect of a Hypocretin/Orexin Antagonist on Neurocognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern California Institute of Research and Education (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas C. Neylan, M.D., Principal Investigator, Northern California Institute of Research and Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NEY-1413
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
Keywords: Sleep Aid
MeSH Terms: interventions — almorexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Almorexant 100mg (Experimental): Subjects will receive a one-time dose of Almorexant 100mg.
  Interventions: Drug: Almorexant
- Almorexant 200mg (Experimental): Subjects will receive a one-time dose of Almorexant 200mg.
  Interventions: Drug: Almorexant
- Zolpidem (Active Comparator): Subjects will receive a one-time dose of Zolpidem 10mg.
  Interventions: Drug: Zolpidem 10mg
- Placebo (Placebo Comparator): Subjects will receive a one-time dose of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Almorexant — 100mg
  Arms: Almorexant 100mg
Drug: Almorexant — 200mg
  Arms: Almorexant 200mg
Drug: Zolpidem 10mg — 10mg
  Other Names: Ambien
  Arms: Zolpidem
Drug: Placebo — One-time dose of Placebo
  Arms: Placebo

SUMMARY:
In recent years, there has been increased focus on cognitive side effects of sleep-inducing medications that may contribute to unusual behavior during unexpected awakenings during the night. Concerns regarding these side effects have led to a class Food and Drug Administration (FDA) warning for all sleep-inducing medications. Almorexant is an experimental sleep-inducing medication in a new class of medications that is being extensively developed by multiple pharmaceutical companies. Medications in this class block wake/arousal centers in the brain that function with proteins called hypocretins. The goal of this study is to evaluate the impact on cognitive performance of almorexant vs. zolpidem (an approved sleep aid) or placebo.

DETAILED DESCRIPTION:
Up to 216 healthy volunteers will be enrolled to participate in the 10 day study. After screening procedures have been completed (at SFVAMC), Days 1 - 7 will take place in subjects' homes, where their sleep/wake activity will be monitored. Days 8 - 10 will take place at Moffitt Hospital. On Day 10, subjects will take one dose of either almorexant 100mg, almorexant 200mg, zolpidem 10mg, or placebo. Cognitive tests will be administered to subjects throughout Day 10. Subjects will return for follow-up safety labs within 5 - 12 days of dosing with study medication. Based on animal studies, it is anticipated that subjects who take almorexant will be less cognitively impaired than those who take zolpidem.

ELIGIBILITY:
To participate in the study, participants must:

* Be between the ages of 19 and 39
* Be in good physical health
* Be a good sleeper with consistent bedtimes and wake times
* Not have problems falling or staying asleep
* Be a non-smoker
* Meet our other study criteria

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2011-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
A comparison between dosing groups on performance on neurocognitive measures | Within a 7-hour window post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Neylan, M.D., Principal Investigator — Northern California Institute of Research and Education
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States